CLINICAL TRIAL: NCT05678283
Title: A Phase 1, 2-Part, Open-label Study to Determine the Absorption, Metabolism, and Elimination of [14C]CC-90010 in Participants With Advanced Solid Tumors
Brief Title: A Study of Absorption, Metabolism, and Elimination CC-90010 in Participants With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA076-001; 2021-005203-13 (EudraCT Number)
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors
Keywords: CC-90010; Neoplasms; Solid Tumors; [14C]CC-90010; BMS-986378; BET Inhibitor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: CC-90010 followed by [14C]CC-90010 (Experimental)
  Interventions: Drug: [14C]CC-90010; Drug: CC-90010
- Part 2: CC-90010 (Experimental)
  Interventions: Drug: CC-90010

INTERVENTIONS:
Drug: [14C]CC-90010 — Specified dose on specified days
  Arms: Part 1: CC-90010 followed by [14C]CC-90010
Drug: CC-90010 — Specified dose on specified days
  Other Names: BMS-986378

SUMMARY:
The purpose of this study is to assess the absorption, metabolism, and elimination of CC-90010 and its metabolites following a single oral dose of radiolabeled CC-90010 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 18 years of age
* Has histological or cytological confirmation of advanced solid tumors including those who have progressed on standard anticancer therapy or for whom no other approved conventional therapy exists
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1

Exclusion Criteria:

* Persistent diarrhea National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade ≥ 2
* History of concurrent second cancers requiring active and ongoing systemic treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-09 (Estimated); Primary Completion 2024-04-29 (Estimated); Study Completion 2024-04-29 (Estimated)

PRIMARY OUTCOMES:
Total [14C]-radioactivity in whole blood, plasma, urine, and feces (and vomit, if applicable) | Up to 26 Days
Cumulative elimination of total [14C]-radioactivity (as a fraction of the radioactive dose) in urine and feces (and vomit, if applicable) | Up to 14 Days
Total [14C]-radioactivity whole blood to plasma ratios | Up to 26 Days
Peak plasma drug concentration (Cmax) | Up to 26 Days
Time to peak plasma drug concentration (Tmax) | Up to 26 Days
Area under the concentration-time curve from time zero to time the time of the last measurable concentration (AUC[0-T]) | Up to 26 Days

SECONDARY OUTCOMES:
Biotransformation of [14C]CC-90010 as [14C]-related metabolites in plasma, urine, and feces | Up to 26 Days
Number of participants with adverse events (AEs) | Up to 26 Months
Number of participants with physical examination abnormalities | Up to 26 Months
Number of participants with vital sign abnormalities | Up to 26 Months
Number of participants with electrocardiogram (ECG) abnormalities | Up to 26 Months
Number of participants with clinical laboratory abnormalities | Up to 26 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0002, Madrid, M, Spain

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html.

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome